CLINICAL TRIAL: NCT01194349
Title: The Role of Reactive Thrombocytosis in Children With Pneumococcal Infection
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Department of Pediatrics, WanFang Hospital, Department of Pediatrics
Other Study IDs: WFH-PED 001, Version 2.990526
Record Dates: First submitted 2010-08-31; First posted 2010-09-03 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-05

CONDITIONS: Thrombocytosis; S. Pneumoniae Infection
Keywords: S. pneumoniae; thrombocytosis; pediatric patients; The study aimed to understand the diagnostic value of thrombocytosis in children with S. pneumoniae infection
MeSH Terms: conditions — Thrombocytosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Thrombocytosis, mostly reactive in nature, is common in pediatric hospitalized patients with infections. Streptococcus pneumoniae (S. Pneumoniae) is the most common pathogen. In this study, the investigators investigated the associations of clinical profiles and thrombocytosis and evaluated platelet counts, leukocyte counts and CRP levels as predictors of hospitalization days in patients with S. pneumoniae infection.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with pneumococcal infection.

Exclusion Criteria:

* Patients with automatic discharge.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric hospitalized patients less than 18 year-old.
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Jinn-Li Wang, Taipei, Taiwan